CLINICAL TRIAL: NCT05177536
Title: Phase 2 Study of Iberdomide Maintenance Therapy Following Autologous Stem Cell Transplant in Patients With Multiple Myeloma
Brief Title: Iberdomide Maintenance Therapy in Patients With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0852-21-FB
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iberdomide (Experimental): Iberdomide will be dosed at 1.0 mg orally daily on days 1-21 of a 28-day cycle
  Interventions: Drug: Iberdomide

INTERVENTIONS:
Drug: Iberdomide — Iberdomide is a novel potent cereblon E3 ligase modulator
  Other Names: cereblon E3 ligase modulator

SUMMARY:
Lenalidomide maintenance therapy following autologous stem cell transplant (ASCT) is standard of care for patients with multiple myeloma. However, nearly all patients will experience disease relapse and lenalidomide's toxicity profile leads to treatment discontinuation in 30% of patients after one year. Iberdomide is a novel potent cereblon E3 ligase modulator with a favorable side effect profile. Investigators hypothesize that iberdomide maintenance therapy may result in at least 80% of subjects completing one year of maintenance.

This study will determine the feasibility, safety and efficacy of iberdomide maintenance therapy post-autologous stem cell transplant (ASCT). Around day 100 after ASCT, patients will be assessed to determine study eligibility. Enrolled participants will take iberdomide pills by mouth on days 1-21 of each 28 day cycle. Physical exams, well-being status and blood and/or urine sampling will be conducted and evaluated before each cycle. Treatment will continue until disease progression or toxicity. Follow-up visits with similar testing will occur every 12 weeks until disease relapse or progression or another treatment for the disease is begun.The results from this study will inform the feasibility of pursuing a study comparing iberdomide to lenalidomide maintenance post-ASCT.

DETAILED DESCRIPTION:
Lenalidomide maintenance therapy following autologous stem cell transplant (ASCT) is standard of care for patients with multiple myeloma. However, nearly all patients will experience disease relapse and lenalidomide's toxicity profile leads to treatment discontinuation in 30% of patients after one year. Iberdomide is a novel potent cereblon E3 ligase modulator with a favorable side effect profile. Investigators hypothesize that iberdomide maintenance therapy may result in at least 80% of subjects completing one year of maintenance.

This is a phase II study to determine the feasibility, safety and efficacy of iberdomide maintenance therapy post-autologous stem cell transplant (ASCT). Around day 100 after ASCT, patients will be assessed to determine study eligibility. Prior to each 28 day cycle, enrolled participants will have health evaluations, well-being assessment and lab tests. Blood and/or urine will be collected for routine tests, disease status and drug effects. Participants will take iberdomide pills by mouth at 1.0 mg PO daily on days 1-21 of each cycle. Treatment will continue until disease progression or toxicity. Participants on study drug at year 1 & 2 will have bone marrow biopsies to assess the disease. Follow-up visits with similar testing will occur every 12 weeks until disease relapse or progression or another treatment for the disease is begun. Study objectives include determination of the proportion of participant completing one year of maintenance treatment, median progression free survival (PFS), minimal residual disease (MRD)-negativity rate at one year post-study drug initiation, sustained MRD-negativity rate, rate of conversion from MRD-positive to negative; overall survival (OS); and safety profile. The results from this study will inform the feasibility of pursuing a phase 3 study comparing iberdomide to lenalidomide maintenance post-ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at consent, ≥19 years old in Nebraska (age of consent)
* Willing and able to provide informed consent to and abide by the protocol
* Documented diagnosis of active measurable Multiple Myeloma (MM):

  * M-protein (serum and/or urine protein electrophoresis (SPEP or UPEP)): SPEP ≥ 0.5 g/dL or UPEP ≥ 200 mg/24 hours and/or
  * Light chain MM without measurable disease in the serum or urine: serum immunoglobulin free light chain ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa-lambda free light chain ratio
* Prior MM therapy

  * Initiation of induction therapy within 12 months of enrollment
  * No prior progression after initial therapy (participants whose induction therapy changed because of suboptimal response or intolerance remain eligible, provided they do not meet criteria for progression as per the 2016 International Myeloma Working Group (IMWG) Response Criteria and no more than two regimens allowed, excluding dexamethasone alone
  * No prior allogeneic hematopoietic stem cell transplant or solid organ transplant
* Autologous Stem Cell Transplant (ASCT) with high dose melphalan (140-200 mg/m2) and in a documented continued partial response or better, per IMWG criteria at 80-110 day post-ASCT
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* All participants must agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment
* All male and female participants must follow all requirements defined in the Pregnancy Prevention Plan in the protocol
* Female participants of childbearing potential (FCBP), achieved menarche at some point; has not undergone a hysterectomy or bilateral oophorectomy and not naturally postmenopausal for at least 24 consecutive months, i.e, has had menses at any time in the preceding 24 consecutive months; (amenorrhea following cancer therapy does not rule out childbearing potential) must:

  * Have two negative serum or urine pregnancy tests as verified by investigators prior to starting study treatment
  * Must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment, even if practicing true abstinence from heterosexual contact
  * Commit to either true abstinence from heterosexual contact (reviewed on a monthly basis and source documented) or agree to use, and to comply with use of two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of iberdomide
* Male participants must:

  * Male participants must practice complete abstinence, acceptable when this aligns with the preferred and usual lifestyle of participant [periodic abstinence (e.g. calendar, ovulation, symptothermal or post-ovulation methods) and withdrawal are not acceptable methods] or agree to use a condom during sexual contact with a pregnant female or a FCBP while taking iberdomide, during dose interruptions and for at least 90 days following the last dose of iberdomide, even if he has undergone a successful vasectomy
  * Must agree to refrain from donating sperm while on study treatment, during dose interruptions and for at least 90 days following last dose of study treatment

Exclusion Criteria:

* Participation in another clinical study with an investigational product within 28 days prior to enrollment
* Female who is pregnant, nursing or breastfeeding, or who intends to become pregnant during study participation
* Any significant medical condition or psychiatric illness that would prevent participation in the study as determined by the treating physician
* Multiple Myeloma (MM) disease progression, as defined by 2016 International Myeloma Working Group (IMWG) Response Criteria following Autologous Stem Cell Transplant (ASCT) prior to enrollment
* Non-secretory MM
* Plasma cell leukemia or light chain amyloidosis
* Any of the following laboratory abnormalities within 14 days of enrollment:

  * Absolute neutrophil count (ANC) < 1,000/μL
  * Platelet count < 75,000/μL
  * Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
  * Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST)or serum glutamic pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≥ 2.0 x upper limit of normal (ULN)
  * Serum total bilirubin and alkaline phosphatase > 1.5 x ULN
  * Serious renal impairment ([CrCl] < 50 mL/min) or requiring dialysis
* Peripheral neuropathy ≥ Grade 2
* Gastrointestinal disease that may significantly alter absorption of iberdomide or inability to take medications by mouth
* Prior history of malignancies, other than MM, unless free of the disease for ≥ 5 years prior to enrollment, excluding:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histological findings of prostate cancer such, e.g., T1a or T1b using Tumor/Node/Metastasis (TNM) classification of malignant tumors or prostate cancer that is curative
* History of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, or pomalidomide
* Received any of the following within 14 days prior to enrollment:

  * Plasmapheresis
  * Major surgery (as defined by investigators
  * Radiation therapy other than local therapy for MM associated bone lesions
  * Use of any systemic myeloma drug therapy
* Any one of the following:

  * Clinically significant abnormal electrocardiogram (ECG) finding within 14 days of enrollment
  * Congestive heart failure (New York Heart Association Class III or IV)
  * Myocardial infarction within 12 months prior to enrollment
  * Unstable or poorly controlled angina pectoris, including the Prinzmetal variant of angina pectoris
* Current or prior use of immunosuppressive medication within 14 days prior to enrollment, excluding:

  * Intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography scan premedication)
* Taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St. John's Wort or related products within two weeks prior to dosing and during the study
* Positive test for human immunodeficiency virus (HIV), chronic or active hepatitis B, or active hepatitis A or C
* Prior therapy with iberdomide
* Unable or unwilling to undergo protocol required thromboembolism prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Able to Complete a Minimum of One Year of Ttherapy | 1 year
  The number of eligible participants who remain on study receiving iberdomide for at least one year without disease progression among all eligible study participants who began protocol treatment will be determined.

SECONDARY OUTCOMES:
Median Progression-free Survival | 5 years
  Progression-free survival (PFS) for all participants will be determined. This defined as the time from enrollment to documentation of disease progression, using 2016 International Myeloma Working Group (IMWG) Response Criteriacriteria, or death without disease progression.
Minimal Residual Disease-negativity Rate at Day 100 | 100 Days
  An estimate of the Minimal Residual Disease (MRD)-negativity rate at day 100 post-initiation of maintenance therapy will be made.
Minimal Residual Disease-negativity Rate at One Year | 1 year
  An estimate of the Minimal Residual Disease (MRD)-negativity rate at one year post-initiation of maintenance therapy will be made.
Minimal Residual Disease-negativity Rate at Two Years | 2 years
  An estimate of the Minimal Residual Disease (MRD)-negativity rate at two years post-initiation of maintenance therapy will be made.
Sustained Minimal Residual Disease-negativity Rate | 1 year
  The sustained Minimal Residual Disease (MRD)-negativity rate, defined as MRD-negativity at study entry and at one year post-initiation of maintenance therapy will be determined.
Rate of Conversion From Minimal Residual Disease-positive to Minimal Residual Disease-negative | 1 year
  The percentage of participants found to be Minimal Residual Disease (MRD) positive at enrollment and MRD negative at one year post-initiation of maintenance therapy among participants meeting the criteria for MRD-positivity at enrollment will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Holstein, MD, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No